CLINICAL TRIAL: NCT02898233
Title: Augmenting Internet-Based Cognitive Behavioral Therapy for Major Depressive Disorder With Low-Level Light Therapy
Acronym: CBT/LLLT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Pilot study was halted due to lack of resources.
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Christopher G. Beevers, Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-09-0100
Record Dates: First submitted 2016-08-24; First posted 2016-09-13 (Estimated); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Depression
Keywords: depression; internet-based; treatment; low-level light therapy; LLLT; deprexis
MeSH Terms: conditions — Depression | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Deprexis and active LLLT (Active Comparator): Participants will have access to Deprexis and will receive active low-level light therapy (4 days X 8 minutes of active LLLT)
  Interventions: Other: Deprexis; Device: Active low-level light therapy
- Deprexis and sham LLLT (Sham Comparator): Participants will have access to Deprexis and will receive sham low-level light therapy (4 days X 5 seconds of active LLLT and 55 seconds of sham LLLT)
  Interventions: Other: Deprexis; Device: Sham low-level light therapy
- Deprexis only (Other): Participants will have access to Deprexis but will not receive real or sham LLLT
  Interventions: Other: Deprexis

INTERVENTIONS:
Other: Deprexis — Deprexis is an experimental internet-based treatment program for depression created by Gaia (Hamburg, Germany).
Device: Active low-level light therapy — Administration of LLLT consists of applying light of a specific wavelength (1064 nanometers) that intersects with the absorption spectrum of cytochrome oxidase, using a laser diode, the high density laser (HD laser; Cell Gen Therapeutics, LLC). Active LLLT includes 4 days, once per week for 4 weeks, during which LLLT is applied to two alternating positions on the participant's right forehead for 8 minutes total.
  Other Names: LLLT
  Arms: Deprexis and active LLLT
Device: Sham low-level light therapy — Administration of LLLT consists of applying light of a specific wavelength (1064 nanometers) that intersects with the absorption spectrum of cytochrome oxidase, using a laser diode, the high density laser (HD laser; Cell Gen Therapeutics, LLC). Sham LLLT includes 4 days, once per week for 4 weeks, during which sham LLLT (5 seconds active, 55 seconds sham) is applied to two alternating positions on the participant's right forehead for 8 minutes total.
  Other Names: LLLT-sham
  Arms: Deprexis and sham LLLT

SUMMARY:
The purpose of this study is to better understand how low-level light therapy (LLLT) can be used to augment the antidepressant effects of Deprexis, an internet-based treatment program for depression, for participants with current major depressive disorder. The researchers will administer active and placebo LLLT to the right forehead of participants who show an improvement of at least 10% in depressive symptoms from baseline after two weeks of Deprexis treatment.

Hypothesis: Participants who receive active LLLT will show a greater reduction of depressive symptoms than participants who receive placebo LLLT.

DETAILED DESCRIPTION:
1. Online screening Following a digital informed consent, all participants will complete a brief online screening questionnaire to determine the severity level of their depression, using the Center for Epidemiological Studies - Depression Scale (CES-D). Initial consent and screening procedures will be conducted online via Research Electronic Data Capture (REDCap), a secure, on-line assessment tool designed to collect self-report questionnaire data for research studies. Participants with a CES-D score of 16 or higher will be eligible to continue with the study. At this initial screening, eligible participants will also provide contact information (name, email address, and phone number) for a follow-up phone screening.
2. Phone screening Following the online screening, eligible participants will complete a phone screening, the Mini International Neuropsychiatric Interview (MINI), conducted by researchers in the Mood Disorders Laboratory. The phone screening will be audio recorded for quality control purposes. Participants will be eligible to continue on in the study if they meet criteria for current Major Depression without any comorbid disorders, excluding anxiety disorders. Next, participants will complete the Colombia-Suicide Severity Rating Scale (C-SSRS) to assess for suicidality. Any participant who endorses suicidal intent, with or without plan, (i.e., items 4 or 5) within the last six months, will be deemed ineligible. Researchers will provide resources to any participant endorsing suicidal ideation, and will contact authorities if necessary. At the end of the phone screening, eligible participants will be scheduled to come into the Mood Disorders Laboratory for their initial study meeting within a week.
3. Initial meeting

   Participants deemed eligible by the online and phone screenings will come into the Mood Disorders Laboratory within a week of their phone screening. The initial meeting will last approximately one hour. The initial meeting will have several objectives:

   First, participants will provide informed consent. Research personnel will provide participants with detailed oral and written description of all study procedures in order to ensure understanding of all components of the study. Participants will provide informed consent for completing the Deprexis program, pre-treatment questionnaires, daily questionnaires, weekly questionnaires, and post-treatment questionnaires. All questionnaires will be accessed online via REDCap.

   Next, participants will complete several pre-treatment questionnaires. Also, researchers will introduce the Deprexis program, and participants will receive an access code that will allow them immediate access to the Deprexis site. Information about the Deprexis program is detailed below.

   Participants will also complete an eye tracking/pupil dilation task during the meeting. Pupil dilation response to emotional stimuli has been shown to be related to depression. In this pupil dilation task, participants will passively view emotional and neutral stimuli (images). More details about the task are below.
4. Pre-treatment questionnaires Participants eligible to take part in the Deprexis program will complete several pre-treatment questionnaires at the initial meeting.
5. Deprexis All Deprexis treatment will be provided via the Deprexis website: http://deprexis.com/. Participants will have access to this website for twelve weeks. They can access this website as often as they would like. The Deprexis program is self-guided, so participants determine how often they access the material (see below for a description of the Deprexis treatment).

   While participants are engaged in the Deprexis treatment program, they will complete the Quick Inventory of Depressive Symptomatology - Self-Report (QIDS-SR) each week, starting with the pre-treatment meeting. This will be automated within the REDCap system and will serve as our primary outcome measure to determine the efficacy of Deprexis in improving depressive symptoms.

   Researchers will monitor the progression of the Deprexis treatment and the QIDS-SR scores for each participant. Participants will be contacted via phone or email as needed to encourage them to continue participating. Participants whose QIDS-SR scores improve by at least 10% from baseline in the first two weeks of Deprexis treatment will be contacted via phone and email to schedule four weekly LLLT sessions in the lab. Participants whose QIDS-SR scores do not improve by 10% from baseline in the first two weeks within the first six weeks of treatment will not be eligible for LLLT, but will continue to have access to the Deprexis program.

   Participants will be scheduled for their initial meeting within 1 week of their phone screening. After the initial meeting, participants will have immediate access to the Deprexis program. During the 12 weeks that participants have access to the Deprexis program, participants will complete the QIDS-SR weekly and may come into the Gonzalez-Lima Lab for LLLT treatment once weekly for four weeks. The maximum amount of time spent in this study for each participant would therefore be 13 weeks.
6. Daily REDCap questionnaires REDCap will automatically send an email to prompt users to answer questions at several times each day during the course of their enrollment in this study. Participants will respond to questions about their mood, stress level, sleep patterns, social interactions, and recent activity. Several times each week, participants will also indicate which, if any, of the Deprexis CBT techniques they have recently used.
7. LLLT Eligible participants will come into the Gonzalez-Lima Lab in Seay 3.304 at their scheduled appointment times. Written informed consent to receive active or placebo LLLT for four sessions will be collected of all lab participants before the first LLLT session. Each session will last approximately twenty minutes. Participants will receive either active or placebo LLLT for eight minutes (procedure described below). Each participant will receive either active LLLT only for all four sessions or sham LLLT only for all four sessions, but not a combination of active and placebo LLLT. Participants will return to the lab at one-week intervals for four weeks. Following each session, participants will be asked if they experienced any perceived side effects (physical or psychological) from the LLLT treatment. In the unlikely event that a participant experiences adverse effects, appropriate measures will be taken to eliminate these effects, and participants will be dismissed from the study if necessary.
8. Post-treatment questionnaires Following completion of the Deprexis treatment, participants will complete several more questionnaires.
9. Location Researchers in the Mood Disorders Laboratory, located in the Liberal Arts Building at The University of Texas at Austin, will administer and assess the participation of each subject in the Deprexis program. Participants will complete the Deprexis treatment online at a location of their choice. Participants who have shown an improvement in depressive symptoms of at least 10% from baseline in the first two weeks of Deprexis treatment will be scheduled to come into the lab for LLLT treatment.

LLLT treatment will be administered in the Gonzalez-Lima Lab, located in Seay 3.304 at The University of Texas at Austin. Participants will come to the lab for four sessions, held approximately one week apart, each of which will last approximately twenty minutes.

Because Deprexis treatment lasts twelve weeks and LLLT lasts four weeks, participants will continue to complete the Deprexis treatment online in the weeks during and after their LLLT sessions. Participants who do not show a 10% improvement in depressive symptoms from baseline in the first two weeks of the Deprexis program will not be eligible to receive LLLT, but will still have access to the Deprexis treatment for the full twelve weeks.

ELIGIBILITY:
Inclusion Criteria:

* ability to speak, read, and understand English fluently
* owns a smartphone and able to receive emails on their phone and access REDCap on a web browser on their phone
* current depressive episode as determined by the Center for Epidemiological Studies - Depression Screening (CES-D) and Mini International Neuropsychiatric Interview (MINI)

Exclusion Criteria:

* serious medical complications, including conditions that change electrical functioning in the brain (e.g., cancer, diabetes, epilepsy, head trauma, history of brain surgery, neurocognitive impairment, stroke, transient ischemic attack)
* comorbid psychiatric disorders, excluding anxiety disorders, as determined by Mini International Neuropsychiatric Interview (MINI)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02; Primary Completion 2020-11 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Self-Report (QIDS-SR) | Week 0 to Week 12, one time per week
  Change in QIDS-SR score from Week 0 to Week 12

SECONDARY OUTCOMES:
Deprexis usage | through study completion; an average of 540 minutes of usage over 12 weeks
  total minutes that participants use Deprexis over 12 weeks
Inventory of Depression and Anxiety Symptoms (IDAS) | Week 0, Week 12
Tridimensional Personality Questionnaire (TPQ) | Week 0, Week 12
Massachusetts General Hospital Antidepressant Treatment Questionnaire (ATRQ) | Week 0, Week 12
Sheehan Disability Scale (SDS) | Week 0, Week 12
Perseverative Thinking Questionnaire (PTQ) | Week 0, Week 12
Questionnaire about daily activities and mood | once per day throughout course of study; daily beginning Week 0 until Week 12
  Brief questionnaire about what the participant did and how the participant felt during the day
Colombia Suicide Severity Rating Scale | through study completion, once during phone screening, thereafter up to once per week, an average of 2 times total
  C-SSRS will be completed at baseline, and up to once per week throughout the study if a participant ever has an increase in suicidal ideation, average of 2 times total

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Beevers, Ph.D., Principal Investigator — Psychology Department, University of Texas at Austin; Francisco Gonzalez-Lima, Ph.D., Principal Investigator — Psychology Department, University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barrett DW, Gonzalez-Lima F. Transcranial infrared laser stimulation produces beneficial cognitive and emotional effects in humans. Neuroscience. 2013 Jan 29;230:13-23. doi: 10.1016/j.neuroscience.2012.11.016. Epub 2012 Nov 27. PMID 23200785
- [Background] Meyer B, Berger T, Caspar F, Beevers CG, Andersson G, Weiss M. Effectiveness of a novel integrative online treatment for depression (Deprexis): randomized controlled trial. J Med Internet Res. 2009 May 11;11(2):e15. doi: 10.2196/jmir.1151. PMID 19632969
- [Background] Schiffer F, Johnston AL, Ravichandran C, Polcari A, Teicher MH, Webb RH, Hamblin MR. Psychological benefits 2 and 4 weeks after a single treatment with near infrared light to the forehead: a pilot study of 10 patients with major depression and anxiety. Behav Brain Funct. 2009 Dec 8;5:46. doi: 10.1186/1744-9081-5-46. PMID 19995444